CLINICAL TRIAL: NCT00383942
Title: The RIPE Study: Ripening Interventions: Prostaglandins vs EASI Catheter
Brief Title: Ripening Interventions: Prostaglandins vs EASI Catheter
Acronym: RIPE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in treatment plan for this population terminated the project
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Scott Graziano, Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109040
Record Dates: First submitted 2006-10-02; First posted 2006-10-04 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Cesarean Section
Keywords: Pregnancy; Extra amniotic saline infusion; Misoprostol; Labor induction
MeSH Terms: interventions — Misoprostol; Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Misoprostol (Active Comparator): Patients randomized to this arm will receive 25 micrograms of misoprostol every four hours.
  Interventions: Drug: Misoprostol
- EASI Catheter (Experimental): Patients randomized to this arm will receive extra amniotic saline infusion (EASI) administered via catheter
  Interventions: Device: Catheter

INTERVENTIONS:
Drug: Misoprostol — Misoprostol,25 micrograms every 4 hours.
  Other Names: Cytotec
  Arms: Misoprostol
Device: Catheter — A catheter with extra amniotic saline infusion (EASI) is placed in the uterus and applies pressure to the cervix to cause it to ripen
  Other Names: EASI
  Arms: EASI Catheter

SUMMARY:
The primary aim of this randomized clinical trial is to compare the effect of misoprostol vs extra amniotic saline infusion via a catheter (EASI) for cervical ripening on the proportion of patients delivered by cesarean section for fetal intolerance of labor versus vaginal delivery. The primary hypothesis is that patients undergoing cervical ripening with EASI catheter are less likely to undergo cesarean section for fetal intolerance of labor when compared to women who receive misoprostol.

DETAILED DESCRIPTION:
Induction of labor is a common obstetrical practice. In fact, the rate of induction has risen to 184/1000 live births. It is well known that a favorable Bishop score, defined as Bishop score 5-8, improves the safety and success rate for induction of labor and vaginal delivery. Several methods for cervical ripening, both mechanical and pharmacological, have been developed to improve Bishop score in women eligible for induction of labor with an unfavorable cervix. These methods include: misoprostol, dinoprostone, intracervical catheter with and without extra-amniotic saline infusion, and laminaria.

Several studies have investigated the optimum cervical ripening agent, and review of current literature supports that misoprostol given in a dose of 25 micrograms every 4 hours intravaginally as the most efficacious and inexpensive regimen while maintaining safe maternal and fetal outcomes. Several studies have shown that misoprostol has a significantly shorter time to delivery compared with other methods of ripening. In fact, in a 2003 Cochrane Database Systematic Review, misoprostol was shown to have increased cervical ripening effectiveness and reduced failure to achieve vaginal delivery in 12-24 hours. Further, while uterine hyper-stimulation and tachysystole were more common in the misoprostol groups, no adverse neonatal outcomes were described. However, misoprostol has been shown to have a higher incidence of cesarean section for fetal intolerance to labor compared to other cervical ripening methods including EASI. Several studies support the ideal route of administration and dosage of misoprostol to be 25 micrograms every 4 hours intravaginally. This regimen leads to effective cervical ripening while reducing the dose-dependent effect of misoprostol on uterine tachysystole and hyperstimulation. Another aspect to consider in cervical ripening method is cost. Misoprostol is much less expensive than other methods including dinoprostone. In fact, one article reports that the average cost per patient for misoprostol treatment was $85 compared to $606 for dinoprostone insert.

Extra-amniotic saline infusion (EASI) has been introduced as a mechanical, non-pharmacological cervical ripening method. It involves placement of a Foley catheter through the cervix and is supplemented with continuous extra-amniotic infusion of saline. This is thought to improve prostaglandin release, resulting in shortened duration of labor. Several studies have been performed to determine the safety and efficacy of the EASI method.

Since misoprostol is efficacious, safe, and inexpensive, it is a superior method for cervical ripening and will act as a control for an experimental group undergoing cervical ripening with the EASI catheter. Our hypothesis is that cervical ripening with the EASI method will result in fewer cesarean sections for fetal intolerance to labor as compared to misoprostol. Furthermore, patients undergoing cervical ripening with EASI will experience a shorter time to delivery, have less expense, have fewer adverse effects, and will be more satisfied with EASI catheter than with misoprostol.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Cephalic presentation
* 36 completed weeks of gestation
* Intact membranes
* Unfavorable cervix (defined as Bishop score < 5)
* Indication for induction of labor
* Fetal Station less than or equal to -3

Exclusion Criteria:

* Clinically significant vaginal bleeding
* Evidence of spontaneous labor (3 contractions in 10 minutes)
* Contraindication to induction of labor or to use of prostaglandins
* Fetal station higher than -3

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-08-31 (Actual); Primary Completion 2008-06-18 (Actual); Study Completion 2008-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Graziano, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data

REFERENCES:
- [Background] Johnson DP, Davis NR, Brown AJ. Risk of cesarean delivery after induction at term in nulliparous women with an unfavorable cervix. Am J Obstet Gynecol. 2003 Jun;188(6):1565-9; discussion 1569-72. doi: 10.1067/mob.2003.458. PMID 12824994
- [Background] Afolabi BB, Oyeneyin OL, Ogedengbe OK. Intravaginal misoprostol versus Foley catheter for cervical ripening and induction of labor. Int J Gynaecol Obstet. 2005 Jun;89(3):263-7. doi: 10.1016/j.ijgo.2005.02.010. Epub 2005 Apr 2. PMID 15919393
- [Background] Karjane NW, Brock EL, Walsh SW. Induction of labor using a foley balloon, with and without extra-amniotic saline infusion. Obstet Gynecol. 2006 Feb;107(2 Pt 1):234-9. doi: 10.1097/01.AOG.0000198629.44186.c8. PMID 16449106
- [Background] Sanchez-Ramos L, Peterson DE, Delke I, Gaudier FL, Kaunitz AM. Labor induction with prostaglandin E1 misoprostol compared with dinoprostone vaginal insert: a randomized trial. Obstet Gynecol. 1998 Mar;91(3):401-5. doi: 10.1016/s0029-7844(97)00673-x. PMID 9491868
- [Background] Garry D, Figueroa R, Kalish RB, Catalano CJ, Maulik D. Randomized controlled trial of vaginal misoprostol versus dinoprostone vaginal insert for labor induction. J Matern Fetal Neonatal Med. 2003 Apr;13(4):254-9. doi: 10.1080/jmf.13.4.254.259. PMID 12854927
- [Background] Adeniji OA, Oladokun A, Olayemi O, Adeniji OI, Odukogbe AA, Ogunbode O, Aimakhu CO, Omigbodun AO, Ilesanmi AO. Pre-induction cervical ripening: transcervical foley catheter versus intravaginal misoprostol. J Obstet Gynaecol. 2005 Feb;25(2):134-9. doi: 10.1080/01443610500040737. PMID 15814391
- [Background] Abramovici D, Goldwasser S, Mabie BC, Mercer BM, Goldwasser R, Sibai BM. A randomized comparison of oral misoprostol versus Foley catheter and oxytocin for induction of labor at term. Am J Obstet Gynecol. 1999 Nov;181(5 Pt 1):1108-12. doi: 10.1016/s0002-9378(99)70090-6. PMID 10561627
- [Background] Hofmeyr GJ, Gulmezoglu AM, Pileggi C. Vaginal misoprostol for cervical ripening and induction of labour. Cochrane Database Syst Rev. 2010 Oct 6;2010(10):CD000941. doi: 10.1002/14651858.CD000941.pub2. PMID 20927722
- [Background] le Roux PA, Olarogun JO, Penny J, Anthony J. Oral and vaginal misoprostol compared with dinoprostone for induction of labor: a randomized controlled trial. Obstet Gynecol. 2002 Feb;99(2):201-5. doi: 10.1016/s0029-7844(01)01681-7. PMID 11814497
- [Background] Guinn DA, Goepfert AR, Christine M, Owen J, Hauth JC. Extra-amniotic saline, laminaria, or prostaglandin E(2) gel for labor induction with unfavorable cervix: a randomized controlled trial. Obstet Gynecol. 2000 Jul;96(1):106-12. doi: 10.1016/s0029-7844(00)00856-5. PMID 10862852
- [Background] Sanchez-Ramos L, Kaunitz AM, Wears RL, Delke I, Gaudier FL. Misoprostol for cervical ripening and labor induction: a meta-analysis. Obstet Gynecol. 1997 Apr;89(4):633-42. doi: 10.1016/S0029-7844(96)00374-2. PMID 9083326
- [Background] Meydanli MM, Caliskan E, Burak F, Narin MA, Atmaca R. Labor induction post-term with 25 micrograms vs. 50 micrograms of intravaginal misoprostol. Int J Gynaecol Obstet. 2003 Jun;81(3):249-55. doi: 10.1016/s0020-7292(03)00042-0. PMID 12767565
- [Background] Has R, Batukan C, Ermis H, Cevher E, Araman A, Kilic G, Ibrahimoglu L. Comparison of 25 and 50 microg vaginally administered misoprostol for preinduction of cervical ripening and labor induction. Gynecol Obstet Invest. 2002;53(1):16-21. doi: 10.1159/000049405. PMID 11803223
- [Background] Diro M, Adra A, Gilles JM, Nassar A, Rodriguez A, Salamat SM, Beydoun SN, O'Sullivan MJ, Yasin SY, Burkett G. A double-blind randomized trial of two dose regimens of misoprostol for cervical ripening and labor induction. J Matern Fetal Med. 1999 May-Jun;8(3):114-8. doi: 10.1002/(SICI)1520-6661(199905/06)8:33.0.CO;2-5. PMID 10338065
- [Background] Sharami SH, Milani F, Zahiri Z, Mansour-Ghanaei F. A randomized trial of prostaglandin E2 gel and extra-amniotic saline infusion with high dose oxytocin for cervical ripening. Med Sci Monit. 2005 Aug;11(8):CR381-6. Epub 2005 Jul 25. PMID 16049380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the trial opened at Loyola University Medical Center (Maywood, IL) on 08/31/2006 and closed on 06/05/2008.
Pre-assignment Details: There are no pre-assignment details
Groups:
- Misoprostol: Patients randomized to this arm receive 25 micrograms of misoprostol every 4 hours.
- EASI: Patients randomized to this arm receive an extra amniotic saline infusion via catheter that is placed in the uterus
Period: Overall Study
Arm/Group | Misoprostol | EASI
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises all patients who were randomized
Groups:
- EASI: Patients randomized to this arm receive extra amniotic saline infusion via a catheter that is placed in the uterus
- Total: Total of all reporting groups
Arm/Group | Misoprostol | EASI | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Women Undergoing Cesarean Section for Fetal Intolerance of Labor
Description: The number of women undergoing cesarean section will be compared between the misoprostol arm and EASI arm. The primary hypothesis is that the odds of receiving a cesarean section is lower among patients assigned to EASI when compared to patients who receive misoprostol.
Time Frame: At time of delivery
Population: No participants are included in this analysis because the trial was terminated prematurely.
Groups:
- EASI: Patients randomized to this arm recieve extra amniotic saline infusion (EASI) via a catheter that is placed in the uterus
Arm/Group | Misoprostol | EASI
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 1 year, 9 months.
Groups:
- Misoprostol: Patients assigned to this arm received 25 micrograms of misoprostol every 4 hours
- EASI: Patients assigned to this arm received extra amniotic saline infusion via a catheter that is placed in the uterus
Arm/Group | Misoprostol | EASI
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Misoprostol (N=40) | EASI (N=40)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial was terminated prematurely due to a department policy change regarding inductions of labor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No